CLINICAL TRIAL: NCT02518750
Title: A Phase II Study Incorporating Panobinostat, Bortezomib and Liposomal Vincristine Into Re-Induction Therapy for Relapsed Pediatric T-Cell Acute Lymphoblastic Leukemia or Lymphoma
Brief Title: Re-Induction Therapy for Relapsed Pediatric T-Cell Acute Lymphoblastic Leukemia or Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSALV; NCI-2015-00935 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-07-16; First posted 2015-08-10 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2018-06

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoma, Non-Hodgkin's; Leukemia, T-Cell; Leukemia, B-Cell
Keywords: Hematopoietic Stem Cell Transplantation; Salvage Regimen; Re-Induction Therapy; Multi-agent chemotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, T-Cell; Leukemia, B-Cell | interventions — Dexamethasone; Calcium Dobesilate; Panobinostat; Vincristine; Mitoxantrone; pegaspargase; Bortezomib; Methotrexate; Mercaptopurine; Cytarabine; nelarabine; Cyclophosphamide; Etoposide; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental): Participants with ALL will receive the following interventions in three treatment blocks:
  * Block A: Dexamethasone, panobinostat, liposomal vincristine, mitoxantrone, peg-asparaginase, bortezomib, intrathecal triples.
  * Block B: High-dose methotrexate, 6-mercaptopurine, intrathecal triples, high-dose cytarabine.
  * Block C: Nelarabine or clofarabine, cyclophosphamide, etoposide.
  Interventions: Drug: Dexamethasone; Drug: Panobinostat; Drug: Liposomal vincristine; Drug: Mitoxantrone; Drug: Peg-asparaginase; Drug: Bortezomib; Drug: Intrathecal Triples; Drug: High-dose methotrexate; Drug: 6-Mercaptopurine; Drug: High-dose cytarabine; Drug: Nelarabine; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Clofarabine

INTERVENTIONS:
Drug: Dexamethasone — Given orally (PO).
  Other Names: Decadron®
Drug: Panobinostat — Given PO.
  Other Names: LBH589
Drug: Liposomal vincristine — For intravenous (IV) use only.
  Other Names: Vincristine sulfate liposome injection; VSLI; Marqibo®
Drug: Mitoxantrone — Given IV.
  Other Names: Novantrone®
Drug: Peg-asparaginase — Given IV or intramuscularly (IM).
  In case of allergy or intolerance to Peg-asparaginase, Erwinia L-asparaginase (Erwinase®) will be used. Erwinia L-asparaginase is given by either IV or IM injection.
  Other Names: Peg-L-asparaginase; Pegaspargase; Oncaspar®
Drug: Bortezomib — Given by IV push over 3 to 5 seconds. For IV use only.
  Other Names: Velcade; MLN341; LDP-341
Drug: Intrathecal Triples — Given IT as ITMHA.
  Other Names: ITMHA; Methotrexate/Hydrocortisone/Cytarabine
Drug: High-dose methotrexate — Given intrathecally (IT) or IV.
  Other Names: HDMTX
Drug: 6-Mercaptopurine — Given PO at consistent time each day.
  Other Names: 6-MP; Purinethol®
Drug: High-dose cytarabine — Given IT or IV.
  Other Names: Ara-C; Cytosar-U®
Drug: Nelarabine — Given IV
  Other Names: Arranon®; Compound 506U78
Drug: Cyclophosphamide — Given IV.
  Other Names: Cytoxan®
Drug: Etoposide — Given IV.
  In case of etoposide reactions, IV etoposide phosphate (Etopophos®) will be used.
  Other Names: VP-16; Vepesid®
Drug: Clofarabine — Given IV.
  Clofarabine will be given instead of nelarabine for patients with B-lymphoblastic leukemia and lymphoma in stratum II.
  Other Names: Clolar™; Clofarex

SUMMARY:
This is a phase-II study to evaluate the efficacy of a salvage regimen in children with relapsed T-cell ALL or lymphoma. Peg-asparaginase, mitoxantrone, intrathecal triples (IT) (intrathecal methotrexate/hydrocortisone/cytarabine) (ITMHA) and dexamethasone are commonly used drugs to treat relapsed or refractory acute lymphocytic leukemia or lymphoma (ALL). In this study, the investigators want to know if adding three drugs called panobinostat, bortezomib and liposomal vincristine (VSLI) to this regimen will result in remission (no signs or symptoms of leukemia or lymphoma).

* Panobinostat has been approved by the FDA for treating adults with multiple myeloma, but it has not been approved for use in children and has not been given together with the other drugs used in this study. It has not been widely studied in children.
* VSLI has been approved by the FDA for adults with relapsed or refractory ALL, but has not yet been approved for treating children with leukemia or lymphoma.
* Bortezomib has been approved by the FDA for treating adults with a cancer called multiple myeloma and adults with relapsed mantle cell lymphoma; it has not been approved for treating children.

PRIMARY OBJECTIVE:

* To estimate the complete remission (CR) rate for patients with T-cell lymphoblastic leukemia and lymphoma in first relapse.

SECONDARY OBJECTIVES:

* To evaluate minimal residual disease (MRD) levels at end of each block of therapy.
* To describe the toxicities of vincristine sulfate liposome injection (VSLI) when used in combination with chemotherapy and bortezomib.

DETAILED DESCRIPTION:
This is a study of re-induction therapy that will comprise of three blocks of multi-agent chemotherapy. CR will be evaluated following each block of therapy. All patients will be candidates for hematopoietic stem cell transplant (HSCT) once they achieve negative minimal residual disease (MRD). If patients cannot proceed to HSCT following Block A, they will continue therapy on Block B and Block C until ready for HSCT.

Three Block Induction:

Block A: approximately 5 weeks

* Dexamethasone 10 mg/m^2/day orally (PO) Days 1-8, 15-22 (Total 16 days)
* Panobinostat 24 mg/m^2/dose PO Day 2,4,6
* Liposomal vincristine (VSLI) 2.25 mg/m^2 no cap intravenously (IV) on Days 7, 14, 21, 28
* Mitoxantrone 10 mg/m^2 IV Day 7,14 (In the absence of peripheral blasts, Day 14 Mitoxantrone will be given if WBC ≥1000 and ANC ≥300)
* Peg-asparaginase 2500 units/m^2 on Days 9,23
* Bortezomib 1.3 mg/m^2 IV Days 16, 19, 23, 26
* Intrathecal Triples (IT) (intrathecal methotrexate/hydrocortisone/cytarabine) (ITMHA) Days 1, 7, 14, 21, 28. Additional ITs on Days 10 and 17 for patients with central nervous system (CNS) 2, 3 or traumatic tap with blasts

Block B: approximately 5 weeks

* High-dose methotrexate 8 g/m^2 IV over 24 hours (will not be given to patients with prior cranial irradiation) Day 1
* 6-mercaptopurine 50 mg/m^2 PO days 1-14
* ITMHA Day 1
* High-dose cytarabine 3 g/m^2 IV every 12 hours (Q12H) Days 15 and 16

Block C: approximately 3 weeks

* Nelarabine 650 mg/m^2/day IV Days 1-5 (Clofarabine 40 mg/m^2/day IV Days 1-5 will be given instead of nelarabine for patients with B-lymphoblastic leukemia and lymphoma in stratum II)
* Cyclophosphamide 300 mg/m^2 IV Days 1-5
* Etoposide 100 mg/m^2/day IV Days 1-5

Response evaluation is performed after the end of each treatment block. All patients should proceed to hematopoietic stem cell transplantation (HSCT) after achieving negative minimal residual disease (MRD) when a suitable donor is identified. Patients could continue on Block B and Block C if not ready for HSCT. If after completion of Block C, MRD is persistently positive, the plan will be discussed with the principal investigator and co-principal investigator and the transplant team. Enrollment on ongoing natural killer (NK) cell studies will be considered. For patients who require a second transplant, HAP3R (another clinical trial at St. Jude Children's Research Hospital) may be an option. Donor will be selected according to institutional practices and transplant regimens will be used according to institutional HSCT protocols and guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have relapsed or refractory acute lymphoblastic leukemia or lymphoma (ALL):

  * Stratum I: T-cell lymphoblastic leukemia or lymphoma in first relapse or refractory to one or two courses of frontline induction therapy.
  * Stratum II: B-cell or T-cell lymphoblastic leukemia or lymphoma in second or third relapse or refractory to 2 or 3 induction or re-induction attempts. Patients with Ph+ ALL must be refractory or relapsed after treatment with regimen that included a tyrosine kinase inhibitor (TKI).
* Relapse in ALL is defined as the reappearance (in a patient who has previously achieved remission) of leukemic blasts in the bone marrow.

  * Should flow cytometric analyses suggest relapse (by the reappearance of a similar immunophenotype to the original leukemia) in the presence of <5% blasts morphologically, a repeat bone marrow test is recommended to confirm relapse.
  * Molecular or genetic relapse is characterized by the reappearance of a cytogenetic or molecular abnormality.
* Age is ≤ 21 years (participant has not yet reached 22nd birthday).
* Able to swallow capsules.
* Karnofsky or Lansky performance score is ≥ 60%. The Lansky performance score should be used for participants < 16 years and the Karnofsky performance score for participants ≥ 16 years.
* Prior therapy:

  * There is no waiting period for participants who relapse while receiving therapy if they are free from side effects attributable to such therapy.
  * Emergent radiation therapy, one dose of intrathecal chemotherapy and up to 7 days of steroids or hydroxyurea are permitted before start of treatment in participants who relapse after completion of frontline therapy. Other circumstances must be cleared by PI or medical designee.
  * At least 90 days have elapsed since bone marrow transplant and participant is off immune suppression for ≥ 2 weeks, if applicable.
* Adequate renal function defined as glomerular filtration rate ≥ 60 cc/min/1.73m^2 or serum creatinine based on age as follows:

  * If age is 1 to 2 years, then maximum serum creatinine (mg/dL) is 0.6 for males or females.
  * If age is 2 to 6 years, then maximum serum creatinine (mg/dL) is 0.8 for males or females.
  * If age is 6 to 10 years, then maximum serum creatinine (mg/dL) is 1 for males or females.
  * If age is 10 to <13 years, then maximum serum creatinine (mg/dL) is 1.2 for males or females.
  * If age is 13 to 16 years, then maximum serum creatinine (mg/dl) is 1.5 for males or 1.4 for females.
  * If age is > 16 years, then maximum serum creatinine (mg/dl) is 1.7 for males or 1.4 for females.
* Adequate hepatic function defined as:

  * Direct bilirubin ≤ 1.4 mg/dL (if total bilirubin > 1.4 mg/dL) AND
  * AST and ALT < 5 x ULN for age.
* Adequate cardiac function defined as shortening fraction of ≥ 27% or ejection fraction ≥ 45%.
* Lymphoma participants without bone marrow involvement must have:

  * Absolute neutrophil count (ANC) >1,000/mm3, AND
  * Platelet count ≥50,000/mm^3 (without transfusion support)
  * NOTE: These criteria are waived for participants with leukemia or lymphoma participants with bone marrow involvement.
* Written, informed consent and assent following Institutional Review Board, NCI, FDA and OHRP guidelines.

Exclusion Criteria:

* Prior histone deacytylases (HDAC), DAC, HSP90 inhibitors or valproic acid for treatment of cancer.
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment.
* Impaired cardiac function or clinically significant cardiac diseases, history of arrhythmia (including ventricular fibrillation or torsade de pointes), bradycardia <50 bpm, screening ECG with prolonged QTc or uncontrolled hypertension.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat.
* Patients with diarrhea > CTCAE grade 2.
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol.
* Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting treatment.
* Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies.
* Patients who have undergone major surgery ≤ 4 weeks prior to starting treatment or who have not recovered from side effects of such therapy.
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis B/C.
* Inability to swallow capsules.
* Active, uncontrolled infection or severe concurrent medical disease, including but not limited to congestive heart failure, cardiac arrhythmias, or psychiatric illness.
* Isolated extramedullary relapse (leukemia) or isolated CNS lymphoma.
* Pregnant or lactating (female participant of childbearing potential must have negative serum or urine pregnancy test required within 7 days prior to start of treatment). Male or female of reproductive potential has agreed to use effective contraception method for duration of study treatment.
* Down syndrome.
* Inability or unwillingness or research participant or legal guardian/representative to give written informed consent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2018-03-11 (Actual); Study Completion 2018-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sima Jeha, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients were recruited between Nov. 2016 and Jan. 2018
Groups:
- Study Paticipants: Participants with ALL will receive the following interventions in three treatment blocks:
  * Block A: Dexamethasone, panobinostat, liposomal vincristine, mitoxantrone, peg-asparaginase, bortezomib, intrathecal triples
  * Block B: High-dose methotrexate, 6-mercaptopurine, intrathecal triples, high-dose cytarabine
  * Block C: Nelarabine or clofarabine, cyclophosphamide, etoposide
Period: Overall Study
Arm/Group | Study Paticipants
Started | 3
Completed | 1
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Participants with ALL will receive the following interventions in three treatment blocks:
  * Block A: Dexamethasone, panobinostat, liposomal vincristine, mitoxantrone, peg-asparaginase, bortezomib, intrathecal triples
  * Block B: High-dose methotrexate, 6-mercaptopurine, intrathecal triples, high-dose cytarabine
  * Block C: Nelarabine or clofarabine, cyclophosphamide, etoposide
Arm/Group | Study Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate
Description: All participants who start re-induction Block A therapy are considered evaluable. Any patient who at any time point achieves CR and goes to transplant is considered as a success; or any patient who successfully reaches the end of block C and achieves/remains in CR is considered a success; all other cases are considered as failure.
Time Frame: At the end of each remission re-induction block C (approximately 13 weeks after start of therapy)
Population: Given the very small enrollment number, no statistical analyses was performed.
Groups:
- Study Paticipants: Participants with ALL will receive the following interventions in three treatment blocks:
  * Block A: Dexamethasone, panobinostat, liposomal vincristine, mitoxantrone, peg-asparaginase, bortezomib, intrathecal triples
  * Block B: High-dose methotrexate, 6-mercaptopurine, intrathecal triples, high-dose cytarabine.
  * Block C: Nelarabine or clofarabine, cyclophosphamide, etoposide
Arm/Group | Study Paticipants
Number analyzed (Participants) | 0

2. Secondary Outcome: Block A Minimal Residual Disease (MRD)
Description: MRD will be studied after each cycle of therapy. MRD is considered as positive (i.e., prevalent) if its level is ≥0.01% for ALL. The prevalence of MRD at end of each cycle is defined as proportion of MRD positives; we will estimate these proportions with point and interval estimates.
Time Frame: At the end of Block A therapy (approximately 5 weeks after start of therapy)
Population: Given the very small enrollment number, no statistical analyses was performed.
Arm/Group | Study Paticipants
Number analyzed (Participants) | 0

3. Secondary Outcome: Block B Minimal Residual Disease (MRD)
Description: as for outcome 2
Time Frame: At the end of Block B therapy (approximately 10 weeks after start of therapy)
Population: No participant received Block B therapy.
Arm/Group | Study Paticipants
Number analyzed (Participants) | 0

4. Secondary Outcome: Block C Minimal Residual Disease (MRD)
Description: as for outcome 2
Time Frame: At the end of Block C therapy (approximately 13 weeks after start of therapy)
Population: No participant received Block C therapy.
Arm/Group | Study Paticipants
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Relevant Toxicities
Description: The toxicities of liposomal vincristine (VSLI) when used in combination with chemotherapy will be evaluated. Proportions (probabilities) of relevant toxicities will be estimated with point and interval estimates.
Time Frame: At the completion of therapy (up to approximately 5 months after the start of therapy)
Population: Given the very small enrollment number, no statistical analyses was performed.
Arm/Group | Study Paticipants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected until either the participant died or up to 30 days after protocol treatment.
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=3)
Sepsis (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (9)
Hypernatremia (Metabolism and nutrition disorders) | 1 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3)
Headache (Nervous system disorders) | 1 (3)
Sepsis (Infections and infestations) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1) — Gamma-glutamyltransferase
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Given the very small enrollment number, no statistical analyses was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT02518750/Prot_SAP_000.pdf